CLINICAL TRIAL: NCT00074334
Title: A Phase I/II Study Of A Recombinant Chimeric Protein Composed Of Transforming Growth Factor (TGF)-a And A Mutated Pseudomonas Exotoxin Termed PE38 (TP-38) In Pediatric Patients With Recurrent Or Progressive Supratentorial High Grade Gliomas
Brief Title: TP-38 Toxin in Treating Young Patients With Recurrent or Progressive Supratentorial High-Grade Glioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug company withdrawal of support for investigational agent in this indication.
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett/PBTC Operations and Biostatistics Center Executive Director, Pediatric Brain Tumor Consortium
Purpose: Treatment
Other Study IDs: CDR0000344416; PBTC-013
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood high-grade cerebral astrocytoma; recurrent childhood cerebral astrocytoma; childhood oligodendroglioma; childhood supratentorial ependymoma; recurrent childhood ependymoma; recurrent childhood brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Familial ependymoma | interventions — transforming growth factor(alpha)-Pseudomonas aeruginosa exotoxin (38)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: TGFa-PE38 immunotoxin
Procedure: conventional surgery

SUMMARY:
RATIONALE: The TP-38 toxin can locate tumor cells and kill them without harming normal cells. Giving TP-38 toxin directly into the tumor may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of TP-38 toxin administered directly into the brain and to see how well it works in treating young patients with recurrent or progressive supratentorial high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Phase I

  * Determine the maximum safe volume rate and maximum tolerated infusion concentration of TGFa-PE38 toxin (TP-38) infused through 2 or 3 catheters in pediatric patients with recurrent or progressive supratentorial high-grade glioma.
  * Describe the toxic effects of this drug in these patients.
* Phase II

  * Estimate the efficacy of this drug, in terms of post-infusion survival, in these patients.

Secondary

* Phase I and II

  * Determine the prevalence of epidermal growth factor receptor (EGFR) expression and phosphorylation (activity) in patients treated with this drug.
  * Correlate EGFR expression with qualitative measures (e.g., histology, grade, and other tumor characteristics) and tumor response, survival, and progression-free survival in patients treated with this drug.
* Phase II Only

  * Estimate the objective response rate in patients treated with this drug.
  * Estimate the progression-free survival of patients treated with this drug.

OUTLINE: This is a dose-escalation, multicenter study. Patients in the phase I portion of the study are stratified according to the number of successfully placed catheters (3 catheters vs 2 catheters). Patients in the phase II portion of the study are stratified according to time of recurrence of high-grade glioma (first vs second or greater) and by surgery extent (surgical resection vs stereotactic biopsy) for those with first recurrence only.

* Phase I: Patients undergo stereotactic biopsy or resection of the tumor followed by intratumoral (or tumor bed) catheter placement for treatment infusion. Within 12-48 hours after intratumoral (or tumor bed) catheter placement, patients receive TGFa-PE38 toxin (TP-38) intratumorally through 2 or 3 catheters over 33 to 124 hours. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients (in each stratum) receive escalating volumes until the maximum safe volume (MSV) is determined. Cohorts of 3-6 patients (in each stratum) receive escalating concentrations at the MSV until the maximum tolerated infusion concentration (MTIC) is determined. The MSV and MTIC are defined as the volume and concentration preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive treatment as in phase I at the MSV and MTIC.

Phase I patients are followed post catheter placement, daily during TP-38 infusion, at 30 days, and then every 2 months for 1 year. Phase II patients will be followed for an additional year.

PROJECTED ACCRUAL: A total of 6-105 patients (6-60 for phase I and 45 for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial malignant glioma

  * Recurrent or progressive disease
* Amenable to gross total resection, clinically indicated partial resection, or biopsy
* Tumor must have a single solid portion at least 1 cm and no greater than 5 cm in maximum diameter

  * No tumor crossing midline

    * Tumors invading the corpus callosum that do not extend beyond to midline or into the contralateral hemisphere allowed
  * No more than 1 focus of tumor
  * No tumors involving the brainstem or cerebellum
  * No tumor dissemination (i.e., subependymal or leptomeningeal)
* Must be on steroids ≥ 3 days prior to surgery
* Must have received prior external beam radiotherapy (tumor dose at least 45 Gy) and completed therapy at least 8 weeks before study entry
* No impending herniation, including midline shift greater than 0.5 cm
* No requirement for immediate palliative treatment

PATIENT CHARACTERISTICS:

Age

* 3 to 21

Performance status

* Karnofsky 60-100% (patients over 16 years of age) OR
* Lansky 60-100% (patients age 16 and under)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3*
* Hemoglobin at least 9 g/dL* NOTE: *Transfusion independent

Hepatic

* ALT and AST less than 2.5 times upper limit of normal (ULN)
* PT and PTT no greater than ULN

Renal

* Creatinine less than 1.5 times normal OR
* Glomerular filtration rate greater than 70 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 30 days after study participation
* No uncontrolled seizures
* No active infection requiring treatment
* No unexplained febrile illness
* No known or suspected allergies to local anesthetics
* No systemic disease or other condition that may be associated with unacceptable anesthetic/operative risk and/or that would preclude study completion
* No other malignancy within the past 5 years except curatively treated carcinoma in situ or basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 8 weeks since prior hematopoietic stem cell transplantation

Chemotherapy

* At least 6 months since prior polifeprosan 20 with carmustine implant (Gliadel® wafer)
* At least 4 weeks since prior cytotoxic chemotherapy (6 weeks for nitrosoureas and 2 weeks for vincristine)
* At least 2 weeks since prior non-cytotoxic chemotherapy
* No other prior intracerebral chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* Concurrent steroids allowed

Radiotherapy

* See Disease Characteristics
* No prior focal radiotherapy (e.g., gamma knife radiosurgery, stereotactic radiosurgery, or brachytherapy)
* No concurrent radiotherapy

Surgery

* Not specified

Other

* Recovered from prior therapy
* At least 4 weeks since prior anticancer investigational agents
* No prior localized antitumor therapy for malignant glioma
* No other concurrent investigational agent
* No other concurrent anticancer (including alternative anticancer medicines/treatment) agent or therapy

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2004-05; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Maximum safe volume rate of TP-38 infused through three catheters (Stratum A) or through two catheters (Stratum B).
Maximum tolerated infusion concentration of TP-38 infused through three catheters (Stratum A) or through two catheters (Stratum B).
Toxicities of TP-38
Post-infusion survival (phase II)

SECONDARY OUTCOMES:
EGFR expression and phosphorylation (activity)
Correlation of EGFR expression with tumor histology, tumor grade, tumor response (phase I and phase II) and survival and progression-free survival (phase II).
Post-infusion progression-free survival (phase II)
Objective response (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Roger J. Packer, MD, Study Chair — Children's National Research Institute
Locations (8):
- United States (8):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas